CLINICAL TRIAL: NCT06001931
Title: Reference Values for Handgrip Strength and Bioimpedance Values in Healthy Turkish Children
Brief Title: Determination of Reference Values for Handgrip Strength and Bioimpedance Values in Healthy Turkish Children
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Aydın, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstanbulPMRTRHChldBioimpedans
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Sarcopenia; Child Development
Keywords: children; muscle strength; bioimpedance
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: handgrip force and bioimpedance values in healthy Turkish children. — Demographic characteristics, calf circumference , Hand grip strength , TANITA BIA analysis

SUMMARY:
In this study, our aim is to determine the reference values for the handgrip force and bioimpedance values in healthy Turkish children.

DETAILED DESCRIPTION:
In this study, our aim is to determine the reference values for the handgrip force and bioimpedance values in healthy Turkish children.

The study was planned as a cross-sectional clinical study. All healthy children studying at Hamdi Akverdi Primary School and Halil Bedii Management Secondary School in the Bakırköy region of Istanbul will be included. The date of birth of the children will be learned. It will be determined in which city in Turkey the population is registered.

TANITA BIA analysis and hand grip strength (with jamar) measured in the dominant hand were planned for all children. In addition, the calf circumference of all children will be measured. Written consent forms will be obtained from the families of the children before the evaluation.

It was planned to include 1500 children in the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy children
* Children under 18
* Turkish children

Exclusion Criteria:

* Children with malignancy or known chronic disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Turkish children
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
handgrip strength | 1 interview day
  Handgrip strength will be measured using a Jamar hand grip dynamometer (Model 5030J1, Sammons Preston Rolyan, Bolingbrook, Illinois, USA). Measurements will be taken 3 times in a sitting position with the elbow flexed to 90° and the wrist in neutral position. The measured maximal grip strength will be recorded as hand grip strength.
calf circumference | 1 interview day
  Calf circumference is an anthropometric measurement that indicates fatfree muscle mass and has been considered by the World Health Organization (WHO) the most sensitive index for evaluating the decrease in muscle mass. Calf circumference will be measured with an elastic band over the subject's right leg, both sitting and standing.
Body Mass Index (BMI) | 1 interview day
  BMI will be calculated as weight (kg) divided by height2 (m2)
Skeletal muscle mass | 1 interview day
  Skeletal muscle mass will be evaluated using a Tanita DC-360 multi-frequency body composition analysis device.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA AYDIN, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Tugba Aydin, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu J, Yan Y, Xi B, Huang G, Mi J; China Child and Adolescent Cardiovascular Health (CCACH) Study Group. Skeletal muscle reference for Chinese children and adolescents. J Cachexia Sarcopenia Muscle. 2019 Feb;10(1):155-164. doi: 10.1002/jcsm.12361. Epub 2018 Nov 30. PMID 30499245
- [Background] McCarthy HD, Samani-Radia D, Jebb SA, Prentice AM. Skeletal muscle mass reference curves for children and adolescents. Pediatr Obes. 2014 Aug;9(4):249-59. doi: 10.1111/j.2047-6310.2013.00168.x. Epub 2013 Jun 18. PMID 23776133
- [Background] Rauch F, Neu CM, Wassmer G, Beck B, Rieger-Wettengl G, Rietschel E, Manz F, Schoenau E. Muscle analysis by measurement of maximal isometric grip force: new reference data and clinical applications in pediatrics. Pediatr Res. 2002 Apr;51(4):505-10. doi: 10.1203/00006450-200204000-00017. PMID 11919337
- [Background] Molenaar HM, Selles RW, Zuidam JM, Willemsen SP, Stam HJ, Hovius SE. Growth diagrams for grip strength in children. Clin Orthop Relat Res. 2010 Jan;468(1):217-23. doi: 10.1007/s11999-009-0881-z. Epub 2009 May 21. PMID 19459024